CLINICAL TRIAL: NCT02049983
Title: Levita Magnetic Grasper Device Safety and Performance Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Levita Magnetics (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LEV-TP-0010; Grant 13IEAT-20911 (Other: CORFO)
Record Dates: First submitted 2014-01-28; First posted 2014-01-30 (Estimated); Results first posted 2024-09-25 (Actual); Last update posted 2024-09-25 (Actual); Status verified 2024-09

CONDITIONS: Benign Gallbladder Disease

ARMS (1):
- Use of Levita Magnetics Grasper (Experimental)
  Interventions: Device: Use of Levita Magnetics Grasper

INTERVENTIONS:
Device: Use of Levita Magnetics Grasper

SUMMARY:
The purpose of this study is to determine the Levita Magnetic Grasper Device Safety and Performance in Laparoscopy.

ELIGIBILITY:
Inclusion Criteria:

* Patient is between 18 and 60 years of age

  * Undergoing elective cholecystectomy due to:
  * Cholelithiasis (Gallbladder stones < 2.5cm in longer measurement (length or width))
  * Gallbladder polyps as assessed by ultrasound
  * Absence of non-correctable coagulopathy (INR < 1.4 or, platelet count of < 50,000/mcl)
  * Patient has a body mass index (BMI) ≤ 35 kg/m2 and over 20
  * Patient, or authorized representative, signs a written Informed Consent form to participate in the study, prior to any study mandated determinations or procedure

Exclusion Criteria:

* Emergency presentation with acute gallbladder disease

  * Pancreatitis
  * Jaundice
  * Scleroatrophic gallbladder as shown by ultrasound
  * Biliary tract stones diagnosed before or during surgery
  * Acute cholecystitis
  * Gallbladder Empyema
  * Ongoing peritoneal dialysis
  * Previous abdominal surgery or laparotomy (presence of any previous upper umbilical incision)
  * Presence of umbilical hernia or previous umbilical hernia
  * American Society of Anesthesiologists (ASA) score of III or IV
  * Patient is undergoing treatment for chronic pain of any origin
  * Significant comorbidities: cardiovascular, neuromuscular, chronic obstructive pulmonary disease, and urological disease (renal failure)
  * Patients with signs of gallbladder perforation diagnosed by ultrasound
  * Suspicion of biliary cancer
  * Patients with severe peritonitis
  * Contraindications to pneumoperitoneum
  * Known allergy to paracetamol or NSAIDs
  * Patients with metallic implants (such as pacemakers, prosthesis, etc)
  * Previously diagnosed or suspected of having a history of choledocholithiasis based on any alterations in plasma hepatic enzymes
  * Has a biliary tract > 7mm in size as determined by ultrasound
  * Has a gallbladder wall thickness that is > 5mm
  * Diabetic Blood coagulation issues
  * Has signs of hepatic endocrinology (i.e: cirrhosis, liver failure, increase in liver enzymes, etc.)
  * History of endoscopic papillotomy (i.e: Preoperative indication of endoscopic retrograde cholangiopancreatography (ERCP)
  * Patient is pregnant or wishes to become pregnant during the length of study participation or lactation
  * Patient is not likely to comply with the follow-up evaluation schedule
  * Patient is participating in a clinical trial of another investigational drug or device
  * Patient is mentally incompetent or a prisoner
  * Known or suspected drug or alcohol abuse
  * Patient has systemic infection or evidence of any surgical site infection (superficial or organ space)
  * Patient has compromised immune system or autoimmune disease (WBC < 4000 or > 20,000), including prior or pending treatment for HIV or Hep. C
  * Patient intra-operatively needs an additional surgery while undergoing elective cholecystectomy

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 50 (Actual)
Dates: Start 2014-01; Primary Completion 2015-03 (Actual); Study Completion 2015-03 (Actual)

CONTACTS AND LOCATIONS:
Locations (3):
- Chile (3):
  - Hospital Luis Tisne, Santiago, Santiago Metropolitan
  - Hospital Padre Hurtado, Santiago, Santiago Metropolitan
  - Hospital Salvador, Santiago, Santiago Metropolitan

REFERENCES:
- [Background] Rivas H, Robles I, Riquelme F, Vivanco M, Jimenez J, Marinkovic B, Uribe M. Magnetic Surgery: Results From First Prospective Clinical Trial in 50 Patients. Ann Surg. 2018 Jan;267(1):88-93. doi: 10.1097/SLA.0000000000002045. PMID 27759614

RESULTS

PARTICIPANT FLOW:
Groups:
- Use of Levita Magnetics Grasper: Use of Levita Magnetics Grasper
Period: Overall Study
Arm/Group | Use of Levita Magnetics Grasper
Started | 50
Completed | 50
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Use of Levita Magnetics Grasper
Number analyzed (Participants) | 50
Age, Continuous [Mean (Standard Deviation); unit: years] | 39 (12.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 45
  Male | 5
Region of Enrollment [Number; unit: participants]
  Chile | 50
BMI [Mean (Standard Deviation); unit: kg/m squared] | 27.0 (3.6)
Indication for surgery [Number; unit: participants]
  Gallbladder stones | 43
  Gallbladder polyps | 7
Ultrasound assessment of gallbladder thickness [Mean (Standard Deviation); unit: mm] | 1.8 (0.5)
Ultrasound assessment of abdominal wall thickness [Mean (Standard Deviation); unit: cm] | 2.6 (0.6)

OUTCOME MEASURES:

1. Primary Outcome: Safety Assessment of AEs
Description: Absence of any damage or side effect to the patient directly produced by the device during the surgery
Time Frame: During surgery
Measure: Count of Participants; unit: Participants
Arm/Group | Use of Levita Magnetics Grasper
Number analyzed (Participants) | 50
Participants
  No device related adverse events | 50
  Device related adverse events | 0

2. Primary Outcome: Feasibility of Mobilization
Description: Ability to adequately mobilize the organ during the surgery
Time Frame: Intra-operative
Measure: Count of Participants; unit: Participants
Arm/Group | Use of Levita Magnetics Grasper
Number analyzed (Participants) | 50
Participants
  Organ adequately mobilized | 50
  Excellent quality of exposure | 45
  Sufficient quality of exposure | 5
  Insufficient quality of exposure | 0

ADVERSE EVENTS:
Time Frame: 30 days
Arm/Group | Use of Levita Magnetics Grasper
All-Cause Mortality (participants affected / at risk) | 0/50
Serious Adverse Events (participants affected / at risk) | 2/50
Other Adverse Events (participants affected / at risk) | 19/50
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Use of Levita Magnetics Grasper (N=50)
hematoma (sub capsular) (Skin and subcutaneous tissue disorders) | 1 (1)
subcutaneous emphysema (Respiratory, thoracic and mediastinal disorders) | 1 (1)
extrahepatic biloma (Gastrointestinal disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Use of Levita Magnetics Grasper (N=50)
petechiae, internal (Skin and subcutaneous tissue disorders) | 19 (19)
petechiae, external (Skin and subcutaneous tissue disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No